CLINICAL TRIAL: NCT04580173
Title: Correlation of Clinical Types and Complexity of Coronary Artery Disease With Patients' Metabolic Profile
Acronym: CorLipid
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: AHEPA University Hospital (Other)
Collaborators: ANALYSIS MEDICAL SA (Unknown); Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Georgios Sianos, Georgios Sianos, Associate Professor of Cardiology MD, PhD, FESC, AHEPA University Hospital, AHEPA University Hospital
Other Study IDs: 95753
Record Dates: First submitted 2020-10-02; First posted 2020-10-08 (Actual); Last update posted 2020-10-12 (Actual); Status verified 2020-10

CONDITIONS: Coronary Artery Disease
Keywords: coronary artery disease; metabolomics
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- SYNTAX score = 0: Patients with nonobstructive CAD (≤50 % diameter stenosis)
  Interventions: Diagnostic Test: metabolomics analysis
- 0 < SYNTAX score <=22: Low SYNTAX group
  Interventions: Diagnostic Test: metabolomics analysis
- 23<=SYNTAX score<=32: Intermediate SYNTAX group
  Interventions: Diagnostic Test: metabolomics analysis
- SYNTAX score>=33: High SYNTAX group
  Interventions: Diagnostic Test: metabolomics analysis

INTERVENTIONS:
Diagnostic Test: metabolomics analysis — Targeted and untargeted metabolomics-based analysis will be performed using Gas Chromatography tandem Mass Spectometry and Liquid Chromatography tandem Mass Spectrometry, in order to quantify serum biomarkers.

SUMMARY:
The purpose of the research project is to investigate the potential association of the complexity and the severity of coronary artery disease (as assessed via SYNTAX score) with patients' metabolic profile. The aim of the study is to combine biochemical, clinical and laboratory data in order to create an algorithm that will enable an individualized therapeutic patient approach.

DETAILED DESCRIPTION:
The objective of this observational study is to expand our knowledge on the biochemical process and pathogenesis of atherogenesis and to recognize clinically important metabolic biomarkers correlated with the severity and clinical presentation of Coronary Artery Disease (CAD). 1050 patients who will undergo coronary angiography will be enrolled in the study. SYNTAX score will be calculated for all participants and their blood samples will be collected before coronary angiography. Metabolomics-based analysis will be performed in order to confirm CAD prognostic biomarkers previously reported in the literature and to investigate their correlations with CAD clinical data. The ultimate aim of this study is to predict the risk of cardiovascular events by incorporating metabolomic information into the SYNTAX score and provide personalized therapeutic guidance to patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients giving voluntary written consent to participate in the study
2. Adults
3. Patients without previous history of coronary artery disease
4. Patients who are admitted in the Department of Cardiology in the AHEPA University General Hospital of Thessaloniki and undergo coronary angiography for clinical purposes

Exclusion Criteria:

1. Cardiac Arrest at admission
2. Patients with serious concurrent disease and life expectancy of < 1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults, of both genders, who are admitted in the Department of Cardiology in the AHEPA University General Hospital of Thessaloniki and undergo coronary angiography for clinical purposes will be studied. Patients with a previous history of coronary artery disease will be excluded. The study includes subjects who 1) have suspected CAD and undergo a scheduled diagnostic angiogram for clinical reasons, and 2) are hospitalized because of an acute coronary syndrome and thus undergo diagnostic angiography (without previous history of CAD).
Sampling Method: Non-Probability Sample
Enrollment: 1050 (Estimated)
Dates: Start 2019-07-12 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Relationship between metabolic profile and the SYNTAX score | 12 months
  Serum metabolomic biomarkers (ceramides, acyl-carnitines, total fatty acids and protein markers: Galectin-3, Neutrophil Gelatinase-Associated Lipocalin, Adiponectin, ApolipoproteinB/ ApolipoproteinΑ-Ι) will be quantified using metabolomics-based methods and enzyme-linked immunosorbent assay. The SYNTAX score will be calculated for all patients. Correlation between patients' metabolic profile and the SYNTAX score will be performed.

SECONDARY OUTCOMES:
Concentration of serum ceramide species | 12 months
  Quantification of serum ceramide species (C18:0/16:0, C18:0/18:0, C18:0/24:0 and C18:0/24:1) using a developed Ultra-high performance liquid chromatography tandem mass spectrometry method.
Concentration of serum acyl-carnitines | 12 months
  Quantification of serum acyl-carnitines (C2, C3, C4, isoC4, C5, isoC5, C6, C8, C10, C12, C14, C16, C18, C18:1 C18:2) using a developed hydrophilic interaction chromatography tandem mass spectrometry method.
Concentration of serum total fatty acids | 12 months
  Quantification of total fatty acids (C10:0, C12:0, C14:0, C15:0, C16:0, C16:1, C17:0, C18:0, C18:1 cis, C18:2 cis, C20:0, C18:3 n6, C18:3 n3, C20:1, C20:2, C22:0, C20:3 n6, C22:1 & C20:4, C23:0, C20:5, C24:0, C24:1, C22:6) using a developed gas chromatography with flame-ionization method.
Concentration of serum selective protein markers | 12 months
  Quantification of selective protein markers (Galectictin-3, NGAL, Adiponectin, ApoB/ ApoΑ-Ι)
Major Adverse Cardiovascular and Cerebrovascular Events | 12 months
  Cardiovascular death, myocardial infarction, stent thrombosis, revascularization and stroke

CONTACTS AND LOCATIONS:
Locations (1):
- AHEPA University Hospital, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: Undecided
The decision to share or not individual participant data with other researchers will depend on the purpose and the scope of the proposed research

REFERENCES:
- [Background] Sianos G, Morel MA, Kappetein AP, Morice MC, Colombo A, Dawkins K, van den Brand M, Van Dyck N, Russell ME, Mohr FW, Serruys PW. The SYNTAX Score: an angiographic tool grading the complexity of coronary artery disease. EuroIntervention. 2005 Aug;1(2):219-27. No abstract available. PMID 19758907
- [Derived] Karagiannidis E, Moysidis DV, Papazoglou AS, Panteris E, Deda O, Stalikas N, Sofidis G, Kartas A, Bekiaridou A, Giannakoulas G, Gika H, Theodoridis G, Sianos G. Prognostic significance of metabolomic biomarkers in patients with diabetes mellitus and coronary artery disease. Cardiovasc Diabetol. 2022 May 7;21(1):70. doi: 10.1186/s12933-022-01494-9. PMID 35525960
- [Derived] Deda O, Panteris E, Meikopoulos T, Begou O, Mouskeftara T, Karagiannidis E, Papazoglou AS, Sianos G, Theodoridis G, Gika H. Correlation of Serum Acylcarnitines with Clinical Presentation and Severity of Coronary Artery Disease. Biomolecules. 2022 Feb 23;12(3):354. doi: 10.3390/biom12030354. PMID 35327546
- [Derived] Karagiannidis E, Sofidis G, Papazoglou AS, Deda O, Panteris E, Moysidis DV, Stalikas N, Kartas A, Papadopoulos A, Stefanopoulos L, Karvounis H, Gika H, Theodoridis G, Sianos G. Correlation of the severity of coronary artery disease with patients' metabolic profile- rationale, design and baseline patient characteristics of the CorLipid trial. BMC Cardiovasc Disord. 2021 Feb 8;21(1):79. doi: 10.1186/s12872-021-01865-2. PMID 33557756